CLINICAL TRIAL: NCT02027896
Title: HIP Fracture Accelerated Surgical TreaTment And Care tracK (HIP ATTACK) Trial
Acronym: HIP ATTACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Population Health Research Institute (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIP ATTACK Trial v5.0
Record Dates: First submitted 2014-01-02; First posted 2014-01-06 (Estimated); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Hip Fractures
Keywords: Perioperative outcomes
MeSH Terms: conditions — Hip Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accelerated medical clearance and surgery (Experimental): Rapid medical clearance with targeted arrival to the operating room within 6 hours of diagnosis of a hip fracture requiring surgical repair.
  Interventions: Other: Accelerated medical clearance and surgery
- Standard surgical care (No Intervention): Surgical hip fracture repair according to the standard timing.

INTERVENTIONS:
Other: Accelerated medical clearance and surgery — Rapid medical clearance with targeted arrival to the operating room within 6 hours of diagnosis of a hip fracture requiring surgical repair.
  Arms: Accelerated medical clearance and surgery

SUMMARY:
HIP ATTACK is an international randomized controlled trial of 3000 patients with a hip fracture that requires a surgical intervention. This trial will determine the effect of accelerated medical clearance and accelerated surgery compared to standard care on the 90-day risk of mortality and major perioperative complication (i.e., a composite of mortality, nonfatal myocardial infarction, nonfatal pulmonary embolism, nonfatal pneumonia, nonfatal sepsis, nonfatal stroke, and nonfatal life-threatening and major bleeding).

ELIGIBILITY:
Inclusion Criteria:

* age ≥45 years; and
* diagnosis of hip fracture during working hours with a low-energy mechanism (i.e., falling from standing height) requiring surgery.

Exclusion Criteria:

* patients requiring emergent surgery or emergent interventions for another reason (e.g., subdural hematoma, abdominal pathology requiring urgent laparotomy, acute limb ischemia, other fractures or trauma requiring emergent surgery, necrotising fasciitis, coronary revascularization, pacemaker-implantation);
* open hip fracture;
* bilateral hip fractures;
* peri-prosthetic fracture;
* therapeutic anticoagulation not induced by a Vitamin K Antagonist, unfractionated heparin, (e.g., administration of therapeutic Low Molecular Weight Heparin (LMWH) (>6,000 u/24h) in the 24 hours prior to enrolment, or intake of any other non-reversible oral anticoagulant(s) for which there is no reversing agent available
* patients on a therapeutic vitamin K antagonist with a history of heparin induced thrombocytopenia (HIT);
* patients refusing participation; or
* patients previously enrolled in the study.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3001 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Composite - major perioperative complication | 90 days
  Composite of mortality, nonfatal myocardial infarction, nonfatal pulmonary embolism, nonfatal pneumonia, nonfatal sepsis, nonfatal stroke, and nonfatal life-threatening and major bleeding
Mortality | 90 days
  All-cause mortality

SECONDARY OUTCOMES:
All-cause mortality | 90 days and 1 year
  Death due to all causes
Vascular mortality | 90 days and 1 year
  Death due to vascular cause
Non-vascular mortality | 90 days and 1 year
  Death due to non-vascular cause
Myocardial infarction | 90 days and 1 year
  Myocardial infarction
Cardiac revascularization procedure | 90 days and 1 year
  i.e., percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG] surgery
New congestive heart failure | 90 days and 1 year
  New congestive heart failure
New clinically important atrial fibrillation | 90 days
  New clinically important atrial fibrillation
Nonfatal cardiac arrest | 30 days and 1 year
  Nonfatal cardiac arrest
Stroke | 90 days and 1 year
  Stroke
Peripheral arterial thrombosis | 90 days and 1 year
  Peripheral arterial thrombosis
Pulmonary embolism | 90 days and 1 year
  Pulmonary embolism
Deep venous thrombosis | 90 days and 1 year
  Deep venous thrombosis
Pneumonia | 90 days and 1 year
  Pneumonia
Sepsis | 90 days and 1 year
  Sepsis
Infection | 90 days
  Infection
Life-threatening bleeding | 90 days
  Life-threatening bleeding
Major bleeding | 90 days
  Major bleeding
New acute renal failure requiring dialysis | 90 days and 1 year
  New acute renal failure requiring dialysis
Peri-prosthetic fracture | 90 days and 1 year
  Peri-prosthetic fracture
Prosthetic hip dislocation | 90 days and 1 year
  Prosthetic hip dislocation
Implant failure | 90 days and 1 year
  Implant failure
Hip re-operation | 30 days and 1 year
  Hip re-operation
Time to first mobilization | 90 days
  Time to first mobilization
Length of hospital stay | 90 days
  Length of hospital stay
Length of critical care stay | 90 days
  Length of critical care stay
Length of rehabilitation stay | 90 days
  Length of rehabilitation stay
New residence in a nursing home | 90 days and 1 year
  New residence in a nursing home
Functional Independence Measure (FIM™) | 30 days and 1 year
  Functional Independence Measure (FIM™)
SF-36 score | 30 days and 1 year
  SF-36 score
Delirium within 7 days of randomization | 7 days
  Delirium within 7 days of randomization
Hospital readmission | 90 days and 1 year
  Hospital readmission
New pressure ulcers | 90 days
  New pressure ulcers
Incisional pain | 30 days
  Incisional pain
Chronic incisional pain | 1 year
  Chronic incisional pain
Acute Kidney Injury | 90 Day
  Acute Kidney Injury
Acute Kidney Injury | 1 Year
  Acute Kidney Injury
Mortality and Institutionalization status of dependents | 30 Days
  Mortality and Institutionalization status of dependents
Mortality and Institutionalization status of dependents | 1 Year
  Mortality and Institutionalization status of dependents
Economic Analysis | 90 Days and 1 Year
  Economic Analysis
Health System Utilization, Long Term Follow up | 2, 5, 10 Years
  Health System Utilization, Long Term Follow up

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Devereaux, MD, PhD, Principal Investigator — McMaster University; Mohit Bhandari, MD, PhD, Principal Investigator — McMaster University
Locations (69):
- United States (5):
  - Regional Medical Center of San Jose, San Jose, California
  - University of Maryland, Baltimore, Maryland
  - Lahey Hospital and Medical Centre, Burlington, Massachusetts
  - Tufts Medical Centre, Washington, Massachusetts
  - Ohio State University Medical Centre, Columbus, Ohio
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (18):
  - South Health Campus, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Concordia Hip and Knee Institute, Winnipeg, Manitoba
  - QEII Health Sciences, Halifax, Nova Scotia
  - Royal Victoria Hospital, Barrie, Ontario
  - Etobicoke General Hospital, Etobicoke, Ontario
  - St. Joseph's Hospital Hamilton, Hamilton, Ontario
  - Hamilton Health Sciences - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Victoria Hospital, London Health Sciences, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Humber River Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Beijing Chaoyang Hospital, Beijing, China
- Fundacion Cardioinfantil, Bogotá, Colombia
- France (2):
  - Centre Hospitalier Lyon Sud, Lyon
  - Nimes University Hospital, Nîmes
- Queen Mary Hospital, High West, Hong Kong
- India (11):
  - Government TD Medical College, Alappuzha
  - Sparsh Hospital, Bangalore
  - PGIMER, Chandigarh
  - Bangalore Baptist Hospital, Hebbāl
  - NH Kolkata, Kolkata
  - CMC Ludhiana, Ludhiana
  - Seven Star Hospital, Nagpur
  - AIIMS Hospital, New Delhi
  - JIPMER, Puducherry
  - Sancheti Institute for Orthopaedics and Rehabilitation, Shivājīnagar
  - Government Medical Hospital, Trivandrum
- Italy (4):
  - Ospedale San Raffaele, Milan
  - Humanitas Research Hospital, Milan
  - IRCCS Galeazzi Orthopedic Institute, Milan
  - ASST Sette Laghi - Ospedale Di, Varese
- Malaysia (2):
  - Hospital Pulau Pinang, George Town
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
- Deventer Ziekenhuis, Deventer, Netherlands
- Pakistan (2):
  - Shifa International Hospitals, Islamabad
  - The Aga Khan University, Karachi
- Poland (3):
  - SPZOZ Szpital Powiatowy w Bochni im M. Wieckiej, Bochnia
  - University Hospital & Educational Center of Medical University in Lodz, Lodz
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej W Myślenicach, Myślenice
- South Africa (3):
  - Groote Schuur Hospital, Cape Town
  - Stellenbosch University, Cape Town
  - Chris Hani Baragwanath Hospital, Johannesburg
- Spain (7):
  - Hospital San Pau, Barcelona
  - Hospital Universitaire Vall d'Hebron, Barcelona
  - Corporació Sanitària Parc Taulí, Barcelona
  - Mutua de Terrassa Hospital, Barcelona
  - Hospital Sant Camil (Consorci Sanitari Garraf), Barcelona
  - Costa del Sol, Marbella
  - Hospital Clinico Universitario de Vallad, Valladolid
- Ramathibodi Hospital, Bangkok, Thailand
- United Kingdom (5):
  - Calderdale & Huddersfield NHS, Huddersfield
  - Chelsea and Westminster Hospital, London
  - West Middlesex Hospital, London
  - Peterborough City Hospital, Peterborough
  - King's Mill Hospital, Sutton in Ashfield

REFERENCES:
- [Derived] Khan JS, Mulazzani F, Devereaux PJ, Bhandari M, Guerra-Farfan E, Patel A, Shanthanna H, Slobogean G, Sigamani A, Umer M, Feibel RJ, Tiboni ME, Tandon V, Harvey V, Balasubramanian K, Vincent J, Tonelli AC, Gilron I, Torrie AM, Borges FK; HIP ATTACK Investigators. Pain as a Driver of Myocardial Injury in Hip Fracture Patients: A Hip Fracture Accelerated Surgical Treatment and Care Track (HIP ATTACK) Trial Secondary Analysis. Anesthesiology. 2026 Feb 1;144(2):289-300. doi: 10.1097/ALN.0000000000005818. Epub 2025 Oct 27. PMID 41147656
- [Derived] HIP ATTACK Investigators. Accelerated surgery versus standard care in hip fracture (HIP ATTACK): an international, randomised, controlled trial. Lancet. 2020 Feb 29;395(10225):698-708. doi: 10.1016/S0140-6736(20)30058-1. Epub 2020 Feb 9. PMID 32050090
- [Derived] Borges FK, Devereaux PJ, Cuerden M, Bhandari M, Guerra-Farfan E, Patel A, Sigamani A, Umer M, Neary J, Tiboni M, Tandon V, Ramokgopa MT, Sancheti P, John B, Lawendy A, Balaguer-Castro M, Jenkinson R, Sleczka P, Nabi Nur A, Wood GCA, Feibel R, McMahon JS, Sigamani A, Biccard BM, Landoni G, Szczeklik W, Wang CY, Tomas-Hernandez J, Abraham V, Vincent J, Harvey V, Pettit S, Sontrop J, Garg AX; HIP ATTACK investigators. Effects of accelerated versus standard care surgery on the risk of acute kidney injury in patients with a hip fracture: a substudy protocol of the hip fracture Accelerated surgical TreaTment And Care tracK (HIP ATTACK) international randomised controlled trial. BMJ Open. 2019 Sep 24;9(9):e033150. doi: 10.1136/bmjopen-2019-033150. PMID 31551393
- [Derived] Borges FK, Bhandari M, Patel A, Avram V, Guerra-Farfan E, Sigamani A, Umer M, Tiboni M, Adili A, Neary J, Tandon V, Sancheti PK, Lawendy A, Jenkinson R, Ramokgopa M, Biccard BM, Szczeklik W, Wang CY, Landoni G, Forget P, Popova E, Wood G, Nabi Nur A, John B, Sleczka P, Feibel RJ, Balaguer-Castro M, Deheshi B, Winemaker M, de Beer J, Kolesar R, Teixidor-Serra J, Tomas-Hernandez J, McGillion M, Shanthanna H, Moppett I, Vincent J, Pettit S, Harvey V, Gauthier L, Alvarado K, Devereaux PJ. Rationale and design of the HIP fracture Accelerated surgical TreaTment And Care tracK (HIP ATTACK) Trial: a protocol for an international randomised controlled trial evaluating early surgery for hip fracture patients. BMJ Open. 2019 May 1;9(4):e028537. doi: 10.1136/bmjopen-2018-028537. PMID 31048449
- See also: HIP ATTACK Pilot Canadian Medical Association Journal (CMAJ) Publication — http://www.cmaj.ca/content/early/2013/11/18/cmaj.130901